CLINICAL TRIAL: NCT03376048
Title: Comparison of Analgesic Efficacy of Local Wound Infiltration Plus Transversus Abdominis Plane Block and Local Wound Infiltration Only After Laparoscopic Colorectal Resection: a Randomized, Double-blind, Non-inferiority Trial
Brief Title: Local Wound Infiltration Plus TAP Block Versus Local Wound Infiltration Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Soo Yeun Park, Colorectal Cancer Center, Kyungpook National University Chilgok Hospital, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNUHC01
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Disorders
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound infiltration plus TAP (Experimental): Wound infiltration placed by surgeon + TAP-LAP placed laparoscopically guided by surgeon
  Interventions: Procedure: Wound infiltration plus TAP
- Wound infiltration (Active Comparator): Wound infiltration placed by surgeon
  Interventions: Procedure: Wound infiltration

INTERVENTIONS:
Procedure: Wound infiltration plus TAP — 1. TAP block: At the beginning of the main surgical procedure the surgeon will perform a TAP with ropivacaine infiltration, bilaterally in the anterior axillary line, between the costal margin and iliac crest in the intermuscular plane between the internal oblique and transversus abdominis muscles, the anesthesiologist under ultrasound guidance, the surgeon under laparoscopic guidance (two "pops" technique).
  2. Wound infiltration : Wound infiltration of ropivacaine will be performed by the surgeon before skin incision.
  Other Names: ropivacaine
  Arms: Wound infiltration plus TAP
Procedure: Wound infiltration — Wound infiltration of ropivacaine will be performed by the surgeon before skin incision.
  Other Names: ropivacaine
  Arms: Wound infiltration

SUMMARY:
The TAP block is typically performed either with ultrasound guidance (TAP-US) or laparoscopic visualization (TAP-LAP): comparison between these two technics showed no differences in pain control and use of opioid analgesics.

The investigators hypothesize that WI is non-inferior to WI + TAP-block with respect to postoperative pain.

DETAILED DESCRIPTION:
In colorectal surgery, laparoscopy and enhanced recovery after surgery (ERAS) programs have significantly improved the short-term outcomes (1). Although the laparoscopic approach reduces pain and recovery time, post-operative pain, nausea and vomiting still represent an issue. In order to reduce opioid related side effects, such as postoperative nausea and vomiting (PONV), constipation and prolonged post-operative ileus, non-opioid based multimodal analgesia have been recently introduced. Although epidural analgesia has gained good success, it does not seem to offer any additional clinical benefits to patients undergoing laparoscopic colorectal surgery compared to alternative analgesic technique within an ERAS program. Both local wound infiltration (WI) and TAP block are common techniques in multimodal postoperative pain treatment, and their association allows to achieve pain control despite a reduced use of opioid analgesics. Furthermore, in a recent single-blind prospective study TAP block resulted superior to wound infiltration alone. The TAP block is typically performed either with ultrasound guidance (TAP-US) or laparoscopic visualization (TAP-LAP): comparison between these two technics showed no differences in pain control and use of opioid analgesics.

The aim of this study is to compare WI + TAP-LAP versus WI alone. The investigators hypothesize that WI is non-inferior to WI + TAP-block with respect to postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years, either sex
* Patients scheduled to undergo elective laparoscopic colorectal surgery under general anesthesia
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Allergies to anesthetic or analgesic medications
* Contraindication to the use of locoregional anesthesia
* Chronic opioid use
* Coagulopathy, Impaired kidney function, uncontrolled diabetes, psychiatric disorders, severe cardiovascular impairment or chronic obstructive lung disease
* Necessity of major resection other than colorectal, palliative surgery
* BMI above 35 kg/m2
* American Society of Anesthesiologists (ASA) physical status above 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Pain numerical rating scale (NRS) | within the first 6 hours after surgery
  1. Pain NRS during rest and cough
  2. NRS scale 0-10: 0, "no pain"; 10, "worst pain imaginable"

SECONDARY OUTCOMES:
Pain NRS | 12, 24, 36, 48, 72 hour after surgery
  1. Pain NRS during rest and cough
  2. NRS scale 0-10: 0, "no pain"; 10, "worst pain imaginable"
Rescue opioid analgesic requirement | postoperative day 0, 1, 2, 3
  Overall postoperative rescue of opioid analgesic requirement described by using the Defined Daily Dose
Postoperative nausea and vomiting scale | 12, 24, 36, 48, 72 hour after surgery
  PONV scores (assessed using a 0 - 2 categorical scale; no nausea/ nausea/ vomiting)
Occurrence of prolonged post-operative ileus | 8 weeks after surgery
  Occurrence of prolonged post-operative ileus (assessed using a 0 - 1 categorical scale; no ileus/ileus)
Time to first oral fluid intake | 8 weeks after surgery
  Time to first oral fluid intake after surgery
Time to first oral soft diet | 8 weeks after surgery
  Time to first oral soft diet after surgery
Length of hospital stay | 8 weeks after surgery
  Length of hospital stay after admission

CONTACTS AND LOCATIONS:
Overall Officials: Soo Yeun Park, MD, Principal Investigator — Kyungpook National University Chilgok Hospital; Corrado Pedrazzani, MD, Principal Investigator — University of Verona Hospital Trust and Colorectal Cancer Center
Locations (2):
- University of Verona Hospital Trust and Colorectal Cancer Center, Verona, Italy
- Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedrazzani C, Park SY, Conti C, Turri G, Park JS, Kim HJ, Polati E, Guglielmi A, Choi GS. Analgesic efficacy of pre-emptive local wound infiltration plus laparoscopic-assisted transversus abdominis plane block versus wound infiltration in patients undergoing laparoscopic colorectal resection: results from a randomized, multicenter, single-blind, non-inferiority trial. Surg Endosc. 2021 Jul;35(7):3329-3338. doi: 10.1007/s00464-020-07771-6. Epub 2020 Jul 6. PMID 32632489
- [Derived] Pedrazzani C, Park SY, Scotton G, Park JS, Kim HJ, Polati E, Guglielmi A, Choi GS. Analgesic efficacy of preemptive local wound infiltration plus laparoscopic-assisted transversus abdominis plane block versus wound infiltration in patients undergoing laparoscopic colorectal resection: study protocol for a randomized, multicenter, single-blind, noninferiority trial. Trials. 2019 Jul 2;20(1):391. doi: 10.1186/s13063-019-3509-y. PMID 31266529